CLINICAL TRIAL: NCT04820803
Title: PILOT CLINICAL TRIAL TO ASSESS THE IMPACT OF ORAL INTERVENTION WITH CETIL PYRIDINIUM CHLORIDE TO REDUCE THE VIRAL LOAD OF SARS-CoV-2
Brief Title: Assessment of the Impact of Oral Intervention With Cetylpyridinium Chloride to Decrease SARS-CoV-2 Viral Load in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosa Tarrago (Other)
Collaborators: Dentaid SL (Industry)
Responsible Party: Sponsor-Investigator, Rosa Tarrago, Principal investigator, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CPC01
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: cetylpyridinium; SARS-CoV-2; COVID-19; mouthwashes
MeSH Terms: conditions — COVID-19 | interventions — Methods; Cetylpyridinium

STUDY DESIGN:
Intervention Model Description: Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 40 subjects in the first group and 40 in the second were required to detect a difference equal to or greater than 5 units. The common standard deviation is assumed to be 10 (12). A loss to follow-up rate of 20% has been estimated.
Who Masked: Participant, Investigator
Masking Description: Randomized double-blind pilot clinical trial (evaluator and patients) in patients with a diagnosis of COVID-19 and symptoms of the disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cetylpyridinium Chloride (CPC) 0,07% (Experimental): patients who rinse with cetylpyiridinium chloride 0,07% mouthwash for 60 seconds
  Interventions: Other: ORAL INTERVENTION WITH CETYLPYRIDINIUM CHLORIDE
- Placebo: Distilled water with the same flavor and coloring as the product to be evaluated (Placebo Comparator): patients who rinse with distilled water mouthwash for 60 seconds
  Interventions: Other: PLACEBO

INTERVENTIONS:
Other: ORAL INTERVENTION WITH CETYLPYRIDINIUM CHLORIDE — one mouthwash containing cetylpyridinium chloride (0.07%) for 60 seconds
  Arms: Cetylpyridinium Chloride (CPC) 0,07%
Other: PLACEBO — one mouthwash containing distilled (placebo) water for 60 seconds
  Arms: Placebo: Distilled water with the same flavor and coloring as the product to be evaluated

SUMMARY:
Pilot, randomized and controlled clinical trial for the evaluation of the decrease in the viral load of SARS-CoV-2 in the oropharynx in patients with COVID-19 through the use of mouthwash containing cetylpyridinium chloride (CPC) (0.07%) in mouthwash.

DETAILED DESCRIPTION:
The objective of the clinical trial is to determine the short-term efficacy of cetylpyridinium chloride (CPC) mouthwashes to assess changes in the threshold cycle value of the analysis of the SARS-CoV-2 oropharyngeal saliva sample, in patients diagnosed with COVID-19 and with symptomatology compatible with the disease. A randomized double-blind pilot clinical trial (evaluator and patients) will be developed in patients with a diagnosis of COVID-19 and symptoms of the disease. The experimental group will perform a single rinse with a mouthwash containing Cetylpyridinium Chloride (CPC) while the placebo group will perform the same rinse, but with a harmless liquid that will act as a placebo. The study will be carried out in the Zaragoza III Health Sector, with patients belonging to the Zaragoza II Health Sector, collaborating with the "Seminario" health center and the Lozano Blesa Clinical University Hospital (HCULB). This project will be carried out in accordance with the CONSORT guidelines for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients older than 18 years and younger than 80 years.
* Patients with a medical indication for a diagnostic test for active infection to SARS-CoV-2
* Patients who present mild symptoms typical of COVID-19 and who have less than three days of evolution
* Patients who have cognitive and motor skills to perform mouthwash correctly.
* Patients who understand and speak Spanish
* Patients who freely give their consent to participate in the study, after a correct understanding of its objectives and procedures.

Exclusion Criteria:

* Patients with hospitalization criteria (moderate or severe symptoms)
* Vulnerable populations such as pregnant, lactating,
* Patients with recent medical diagnosis (≤ 1 month) of pneumonia
* Patients with hyposialia
* Patients with consumption of oral antiseptics (in the form of mouthwash containing CPC, povidone iodine rinses, alcohol mouthwash and essential oils) and toothpastes with CPC during the last month.
* Patients with cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Threshold cycle value of SARS-CoV-2 by Polymerase Chain Reaction (PCR) in saliva samples | 3 months
  Threshold cycle value of SARS-CoV-2 by Polymerase Chain Reaction (PCR) in saliva samples before antd 2hours after mouthwashes
SARS-CoV-2 Nucleocapsid protein in saliva by ELISA | 3 months
  Quantitative determination of SARS-CoV-2 Nucleocapsid protein in saliva by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Seminario Health Center and Lozano Blesa University Clinical Hospital, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No